CLINICAL TRIAL: NCT01215045
Title: Visual Performance of Bilateral AcrySof ReSTOR Aspheric +4
Status: Completed | Type: Observational
Sponsor: Alcon Research (Industry)
Responsible Party: Rick Potvin, Alcon
Other Study IDs: M07-004
Record Dates: First submitted 2008-08-12; First posted 2010-10-05 (Estimated); Last update posted 2010-10-05 (Estimated); Status verified 2010-10

CONDITIONS: Cataract
Keywords: AcrySof ReSTOR Aspheric +4
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ReSTOR +4: AcrySof ReSTOR Aspheric +4
  Interventions: Device: AcrySof ReSTOR Aspheric +4

INTERVENTIONS:
Device: AcrySof ReSTOR Aspheric +4 — Implantation with the AcrySof ReSTOR Aspheric +4 Multifocal Intraocular Lens (IOL)

SUMMARY:
Determine the clinical visual outcomes following bilateral implantation of the AcrySof ReSTOR Aspheric Intraocular Lens (IOL) and to demonstrate what percentage of the subjects obtain spectacle freedom.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with cataracts

Exclusion Criteria:

* Preexisting conditions confounding results; > 1 Diopter preoperative astigmatism

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study participants taken from physician's patient pool implanted with the AcrySof ReSTOR +4 Intraocular Lens (IOL)
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2007-06; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Visual Acuity | 6 months

SECONDARY OUTCOMES:
Contrast sensitivity, patient survey | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Contact Alcon Call Center for Trial Locations, Fort Worth, Texas, United States